CLINICAL TRIAL: NCT02077764
Title: The GRAFT Study: Evaluation of Graft Function, Rejection and Cardiac Allograft Vasculopathy in First Heart Transplant Recipients.
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Tor Skibsted Clemmensen, M.D., PhD student, Aarhus University Hospital Skejby
Other Study IDs: Sagsnr. 1-10-72-153-13; The GRAFT study: Evaluation of (Registry Identifier: GRAFT: Evaluation of Graft function, Rejection and cardiac Allograft vasculopathy in First heart Transplant recipients)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Heart Transplant Recipients
Keywords: heart transplantation,; rejection; cardiac vasculopathy; optical coherence tomography; speckle tracking; Positron Emission Tomography .; exercise capacity
MeSH Terms: conditions — Rejection, Psychology | interventions — Exercise Test; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — At each visit blood samples are taken. These will include:
  1 x 10 ml EDTA-blood
  1 x 10 ml Lithiumheparin-blood
  1 x 10ml Koagel -blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls, healthy individuals: controls
  Interventions: Procedure: Echocardiography
- Heart transplanted patients: Patients
  Interventions: Procedure: OCT and coronary angiography; Procedure: Right heart cat.; Radiation: PET; Procedure: Echocardiography; Procedure: exercise test; Other: blood samples

INTERVENTIONS:
Procedure: OCT and coronary angiography
  Groups: Heart transplanted patients
Procedure: Right heart cat.
  Groups: Heart transplanted patients
Radiation: PET
  Groups: Heart transplanted patients
Procedure: Echocardiography
Procedure: exercise test
  Groups: Heart transplanted patients
Other: blood samples
  Groups: Heart transplanted patients

SUMMARY:
Objective:

* To assess the relationship between coronary allograft vasculopathy (CAV) and graft function, and to evaluate non-invasive methods for CAV diagnosis.
* To assess left ventricular (LV) and right ventricular (RV) function in the acute phase and serially during the first year after transplantation.
* To evaluate the impact of acute and repetitive rejection on the longitudinal myocardial function Hypothesis

  1. Timing of development and degree of CAV can be measured non-invasively combining myocardial longitudinal deformation (by advanced echocardiography) and coronary flow velocity reserve (CFVR) (by echocardiography and PET). This combination of methods can detect CAV before it is angiographically visual and gives supplementary information of the impact on myocardial graft function.
  2. Longitudinal deformation, 3D echocardiography, cardiac magnetic resonance imaging (CMRI) and PET can be used for RV and LV myocardial function assessment and represent more valid markers of the function than standard echocardiography in heart transplant (HTX) patients.
  3. Myocardial longitudinal deformation is a better marker of acute rejections than conventional ejection fraction (EF).

Background The most frequent heart related death causes after HTX are CAV, acute graft failure and rejection.

CAV is characterized by diffuse concentric intima thickening involving both epicardial vessels and the coronary microvascular system. In our clinical approach HTX-patients are followed with annual CAG and standard echocardiography with estimation of LV systolic function by EF. Standard echocardiography has not proven benefit in the diagnosis of CAV. CAG often misses CAV in early phases.

In various cardiac diseases it is well known that ischemia and fibrosis often affect the endocardial longitudinal oriented layers. Longitudinal deformation by advanced echocardiography has shown to be better markers for systolic function in HTX patients compared to standard EF. Longitudinal LV systolic function is dependent of endocardial perfusion. CFVR represents the capacity of the coronary circulation to dilate due to metabolic demands and has been shown to correlate with longitudinal deformation in myocardial infarction. CFVR measurements in HTX patients with advanced echocardiography and PET scan have shown a significant correlation to CAV.

RV failure is an early, potentially fatal, complication to HTX. The function and change over time of RV have not been fully studied using modern echocardiographic techniques or assessment by CMRI.

Acute rejection is an inflammatory response often diagnosed by routine biopsies (gold standard). These are expensive, time consuming and inconvenient for the patient. The role of conventional echocardiography has not yet found a significant role in the diagnostics of acute rejections and furthermore how repeated rejections influence on graft function is not well described.

Study 1 A cross sectional study consisting of 50 stabile HTX patients. These will be selected with 25 patients with no or light CAV and 25 patients with moderate or severe CAV.

Severity of CAV will be evaluated by:

* CAG
* CFVR measurement by advanced echocardiography and PET.

Graft function will be evaluated by:

* Advanced echocardiography at rest end during bicycle exercise.
* CMRI including assessment of LV and RV EF, strain and mass.
* During rest and bicycle exercise echocardiography simultaneously right heart catheterization are performed for hemodynamic measurement

Study 2 A prospective cohort study with 20-25 newly transplanted patients over a period of 12 months.

LV and RV function will be measured by:

* Advanced echocardiography
* CFVR measurement (echocardiography and PET)
* CMRI for LV and RV EF, strain and mass
* Right heart catheterization

Study 3 Prospective examination of correlation between graft function, CAV and rejection. Information of former episodes of acute rejection is collected retrospective. Study objectives are all living HTX patients (approx. 200) in the period of 2011-2013.

Advanced echocardiography (including longitudinal deformation), biopsies (rejection evaluation) and CAG (CAV evaluation).

DETAILED DESCRIPTION:
Objective

1. To assess the relationship between myocardial perfusion, coronary anatomy and longitudinal myocardial function in heart transplanted (HTX) patients with and without coronary allograft vasculopathy (CAV).
2. Evaluation of systolic and diastolic capacity during exercise in HTX patients with and without CAV.
3. Evaluation of non-invasive methods for CAV diagnosis.
4. To assess left ventricular (LV) and right ventricular (RV) function in the acute phase and during follow-up (5 times) the first year after transplantation and furthermore to compare advanced echocardiographic evaluation of graft function with cardiac magnetic resonance imaging (CMRI), right heart catheterization, and positron emission tomography (PET).
5. Finally, to evaluate the impact of acute and repetitive rejection on myocardial graft function measured by standard 2D echocardiography and advanced echocardiography with analysis of longitudinal myocardial function.

Hypothesis

1. Timing of development and degree of CAV can be measured non-invasively combining myocardial longitudinal deformation measurement by advanced echocardiography and coronary flow velocity reserve (CFVR) by echocardiography and PET. This combination of methods can detect CAV before it is angiographic visual and gives supplementary information of the impact on myocardial graft function. This setup might be more appropriate in evaluation of the myocardial graft function and CAV than standard echocardiography and coronary angiography (CAG). Optical coherence tomography (OCT) can detect CAV in early phases and gives supplementary characterization of the plaque.
2. Modern non-invasive methods (longitudinal deformation, 3D echocardiography, CMRI and PET) can be used in RV and LV myocardial function assessment and represents more valid markers of the function than standard echocardiography in HTX patients.
3. During exercise patients with CAV will show impaired longitudinal myocardial deformation and restrictive filling with significant increasing LV and RV filling pressures.
4. Myocardial longitudinal deformation is a better marker of acute rejections than conventional ejection fraction (EF). After an episode of severe acute rejection the graft function will improve, but instances of repetitive rejections will lead to impaired longitudinal systolic function with preserved LV EF.

Background Mean survival after HTX at our center is 15.6 years. Complications remain frequent and serious. In the first postoperative year the main causes of death are graft failure, rejections and infection. At long term follow up main causes of death are CAV and malignancies.

CAV is characterized by diffuse concentric intima thickening involving both epicardial vessels and the coronary microvascular system. After 10 years more than 50% of patients shows angiographic signs of CAV.

In our clinical approach HTX-patients are followed with annual CAG and standard echocardiography with estimation of LV systolic function by EF. EF is often within normal range even though CAV lesions are evident by CAG, suggesting that LV EF is an inappropriate parameter for detecting impaired myocardial function in CAV. Symptoms of graft dysfunction first present themself with severe CAV. Studies have shown that CAG often misses CAV in early phases. OCT is a novel intravascular imaging modality with excellent spatial resolution. It has been used in a few small cross sectional studies with HTX patients and seems like a promising tool for detecting CAV and gives supplementary characterization of the plaque.

In various cardiac diseases it is well known that ischemia and fibrosis often affect the endocardial longitudinal oriented layers leading to abnormal systolic function of both LV and RV. Longitudinal deformation by tissue Doppler and strain analysis has shown to be better markers for systolic function in HTX patients compared to standard measurements such as LV EF. Longitudinal LV systolic function is dependent of endocardial perfusion. CFVR represents the capacity of the coronary circulation to dilate, due to increased myocardial metabolic demands and is expressed by the difference between the hyperaemic and resting flow. CFVR has been shown to correlate with the degree of decreased longitudinal deformation in myocardial infarction. CFVR measurements in HTX patients with color Doppler echocardiography and PET scan have shown a significant correlation to CAV.

RV failure is an early, potentially fatal, complication to HTX. Standard echocardiographic measurement does not seem to reflect the overall RV systolic performance and clinical status of the patient. Prior studies have found impaired RV function after HTX, but most studies of RV function were not performed with simultaneous right heart catheterization or assessment of RV EF by CMRI (golden standard). Overall the function and change over time of RV have not been fully studied using modern echocardiographic techniques or assessment by CMRI.

Acute rejection is an inflammatory response most frequently in the first 6 months after HTX. Two thirds experience rejection episodes within first year.

Rejections are often asymptomatic and associated with poor outcome, including development of CAV. Patients are followed with routine biopsies (gold standard), but these are expensive, time consuming and inconvenient for the patient. The role of conventional echocardiography has not yet found a significant role in the diagnostics of acute rejections and furthermore how repeated rejections influence on graft function is not well described.

Study objective, design and methods Study 1 Design: A cross sectional study consisting of 50 stabile HTX patients. These will be selected with 25 patients with no or light CAV and 25 patients with moderate or severe CAV. 25 matched controls.

Methods:

Severity of CAV will be evaluated by:

* CAG supplied with OCT.
* CFVR measurement by echocardiography with adenosine induced hyperemia.
* CFVR measurement with H215O-PET.

Graft function will be evaluated by:

* 2D and 3D echocardiography (including longitudinal deformation and tissue Doppler)
* Diastolic (and systolic) stress test: Bicycle exercise with simultaneously echocardiography and right heart catheterization.

Blood samples are taken for analysis of myocardial fibrosis markers, CRP, TNT and NT-proBNP.

Study 2 Design: A prospective cohort study with 20 newly transplanted patients over a period of 12 months.

Methods: LV and RV function shall be measured by:

* 2D and 3D echocardiography (including longitudinal deformation, tissue Doppler, CFVR, LV and RV EF),
* CMRI for LV and RV EF, strain and mass
* Right heart catheterization
* H215O-PET at baseline and after 3 month in the assessment of RV function
* Coronary angiography after 3 and 12 month will be supplied with OCT for early signs of CAV development.

Biopsies are performed according to routine protocol after transplantation. Blood samples for analysis of myocardial fibrosis markers, CRP, TNT and NT-proBNP.

Study 3 Design: Prospective examination of correlation between graft function, CAV and rejection. Information of former episodes of acute rejection is collected retrospective. Study objectives are all living HTX patients (approx. 200) in the period of 2011-2013.

Methods: Advanced echocardiography (including longitudinal deformation and tissue Doppler), biopsies (rejection evaluation) and CAG (CAV evaluation).

Publication Plan:

Positive as well as negative result from study 1-3 will be published. We aim at publishing study 1-3 in peer review international, scientific journals. Study 3 is expected to be published in 2014 and study 1 and 2 in 2016. MD, PhD student Tor Skibsted Clemmensen will draft the manuscripts and be 1st author hereof.

Ethical considerations Adenosine, used for CFVR measurement and PET, often causes mild facial flushing, chest discomfort and dyspnoea. After suspended infusion symptoms last less than one minute since half time is below 10 seconds.

Right heart catheterisation is part of the standard protocol after HTX. Only patients in study 1 might be subjected to more catheterisations than normally. Complications are rare with experienced operators.

The radiation dose of H215O-PET is 2-2,5 mSv, approximately the same as one year background radiation. Patients in study 1 will be subjected to one examination, patients in study 2 two examinations.

No additional CAG are made in the studies. OCT examination is considered very safe with a risk of complication <0,5%.

The investigators are convinced that the possible risks are outweighed by the expected benefits from this study and no study-related examinations will be conducted until informed consent form has been signed.

Regional Scientific Ethical Committee of Central Denmark has approve the studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100
* Informed and signed consent

Exclusion Criteria:

* - Coronary stenosis within the first 3 mounts after HTX (donor transmitted coronary atherosclerosis).
* Severe asthma or COLD with FEV1 < 50%
* 2° or 3° AV block
* Pregnancy
* S-creatinine >200 µmol/l
* Allergy towards the contrast agent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Design: A cross sectional study consisting of 50 stabile HTX patients. These will be selected with 25 patients with no or light CAV and 25 patients with moderate or severe CAV. 25 matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Coronary flow velocity reserve | September 2013 to January 2016
  Assessed by tissue Doppler echocardiography and H215O-PET
pulmonary capillary wedge pressure | September 2013 to January 2016
  At rest and during exercise
global longitudinal strain | September 2013 to January 2016
  At rest and during exercise
cardiac allograft vasculopathy | September 2013 to January 2016
  Assessed by coronary angiography and optical coherence tomography

SECONDARY OUTCOMES:
RV-EF | September 2013 to January 2016
  3D echocardiography
Quality of life | September 2013 to January 2016
  Minnesota quality of life questionnaires
CRP, TNT, Nt-ProBNP and fibrosis markers | September 2013 to January 2016
  Correlation between cardiac allograft vasculopathy and biomarkers
tissue Doppler | September 2013 to January 2016
  Correlation between rejection, vasculopathy and tissue Doppler echocardiography- in rest and during exercise
Cardiac output | September 2013 to January 2016
  At rest and during exercise in a HTX population
intima/media radio | September 2013 to January 2016
  Assessed by optical coherence tomography

OTHER OUTCOMES:
Correlation between Rubidium and H2O PET | May 2014 to January 2016
  Patients will be subjected to tests with bodt tracers to validate rubidium as tracer in a HTX population
3D echocardiography as a tool to diagnose vasculopathy | September 2013 to January 2016

CONTACTS AND LOCATIONS:
Overall Officials: Steen H Poulsen, M.D. DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Aarhus N, Denmark

REFERENCES:
- [Background] Clemmensen TS, Munk K, Tram EM, Ilkjaer LB, Severinsen IK, Eiskjaer H. Twenty years' experience at the Heart Transplant Center, Aarhus University Hospital, Skejby, Denmark. Scand Cardiovasc J. 2013 Dec;47(6):322-8. doi: 10.3109/14017431.2013.845688. Epub 2013 Oct 16. PMID 24131212
- [Background] Stehlik J, Edwards LB, Kucheryavaya AY, Benden C, Christie JD, Dipchand AI, Dobbels F, Kirk R, Rahmel AO, Hertz MI; International Society of Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: 29th official adult heart transplant report--2012. J Heart Lung Transplant. 2012 Oct;31(10):1052-64. doi: 10.1016/j.healun.2012.08.002. No abstract available. PMID 22975095
- [Background] Sipahi I, Starling RC. Cardiac allograft vasculopathy: an update. Heart Fail Clin. 2007 Jan;3(1):87-95. doi: 10.1016/j.hfc.2007.02.007. PMID 17545012
- [Background] Tona F, Osto E, Tarantini G, Gambino A, Cavallin F, Feltrin G, Montisci R, Caforio AL, Gerosa G, Iliceto S. Coronary flow reserve by transthoracic echocardiography predicts epicardial intimal thickening in cardiac allograft vasculopathy. Am J Transplant. 2010 Jul;10(7):1668-76. doi: 10.1111/j.1600-6143.2010.03160.x. PMID 20642688
- [Background] Khandhar SJ, Yamamoto H, Teuteberg JJ, Shullo MA, Bezerra HG, Costa MA, Selzer F, Lee JS, Marroquin OC, McNamara DM, Mulukutla SR, Toma C. Optical coherence tomography for characterization of cardiac allograft vasculopathy after heart transplantation (OCTCAV study). J Heart Lung Transplant. 2013 Jun;32(6):596-602. doi: 10.1016/j.healun.2013.02.005. Epub 2013 Mar 15. PMID 23499356
- [Background] Syeda B, Hofer P, Pichler P, Vertesich M, Bergler-Klein J, Roedler S, Mahr S, Goliasch G, Zuckermann A, Binder T. Two-dimensional speckle-tracking strain echocardiography in long-term heart transplant patients: a study comparing deformation parameters and ejection fraction derived from echocardiography and multislice computed tomography. Eur J Echocardiogr. 2011 Jul;12(7):490-6. doi: 10.1093/ejechocard/jer064. Epub 2011 Jun 2. PMID 21636605
- [Background] Logstrup BB, Hofsten DE, Christophersen TB, Moller JE, Botker HE, Pellikka PA, Egstrup K. Correlation between left ventricular global and regional longitudinal systolic strain and impaired microcirculation in patients with acute myocardial infarction. Echocardiography. 2012 Nov;29(10):1181-90. doi: 10.1111/j.1540-8175.2012.01784.x. Epub 2012 Aug 3. PMID 22862151
- [Background] Wu YW, Chen YH, Wang SS, Jui HY, Yen RF, Tzen KY, Chen MF, Lee CM. PET assessment of myocardial perfusion reserve inversely correlates with intravascular ultrasound findings in angiographically normal cardiac transplant recipients. J Nucl Med. 2010 Jun;51(6):906-12. doi: 10.2967/jnumed.109.073833. Epub 2010 May 19. PMID 20484427
- [Background] Fyfe DA, Mahle WT, Kanter KR, Wu G, Vincent RN, Ketchum DL. Reduction of tricuspid annular doppler tissue velocities in pediatric heart transplant patients. J Heart Lung Transplant. 2003 May;22(5):553-9. doi: 10.1016/s1053-2498(02)00653-8. PMID 12742418
- [Background] Goland S, Siegel RJ, Burton K, De Robertis MA, Rafique A, Schwarz E, Zivari K, Mirocha J, Trento A, Czer LS. Changes in left and right ventricular function of donor hearts during the first year after heart transplantation. Heart. 2011 Oct;97(20):1681-6. doi: 10.1136/hrt.2010.220871. Epub 2011 May 17. PMID 21586422
- [Background] D'Andrea A, Riegler L, Nunziata L, Scarafile R, Gravino R, Salerno G, Amarelli C, Maiello C, Limongelli G, Di Salvo G, Caso P, Bossone E, Calabro R, Pacileo G, Russo MG. Right heart morphology and function in heart transplantation recipients. J Cardiovasc Med (Hagerstown). 2013 Sep;14(9):648-58. doi: 10.2459/JCM.0b013e32835ec634. PMID 23442808
- [Derived] Clemmensen TS, Holm NR, Eiskjaer H, Logstrup BB, Christiansen EH, Dijkstra J, Barkholt TO, Terkelsen CJ, Maeng M, Poulsen SH. Layered Fibrotic Plaques Are the Predominant Component in Cardiac Allograft Vasculopathy: Systematic Findings and Risk Stratification by OCT. JACC Cardiovasc Imaging. 2017 Jul;10(7):773-784. doi: 10.1016/j.jcmg.2016.10.021. Epub 2017 Mar 15. PMID 28330670
- [Derived] Clemmensen TS, Eiskjaer H, Logstrup BB, Mellemkjaer S, Andersen MJ, Tolbod LP, Harms HJ, Poulsen SH. Clinical features, exercise hemodynamics, and determinants of left ventricular elevated filling pressure in heart-transplanted patients. Transpl Int. 2016 Feb;29(2):196-206. doi: 10.1111/tri.12690. Epub 2015 Oct 5. PMID 26369751